CLINICAL TRIAL: NCT01684280
Title: Searching for the Most Influential Obesity-related Diabetic Genes and Exploring the Expression Profiles of Those Genes in Taiwanese Undergoing Weight Loss
Brief Title: Obesity-related Genes in Taiwanese Undergoing Weight Loss
Status: Completed | Type: Observational
Sponsor: Sung Ling Yeh (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor-Investigator, Sung Ling Yeh, professor, Taipei Medical University Hospital
Organization: Taipei Medical University Hospital (Other)
Other Study IDs: CRC-06-09-10
Record Dates: First submitted 2012-09-10; First posted 2012-09-12 (Estimated); Last update posted 2012-09-13 (Estimated); Status verified 2012-09

CONDITIONS: Morbid Obesity
Keywords: abdominal adipose tissue; microRNA
MeSH Terms: conditions — Obesity, Morbid | interventions — Sex

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — Paired samples of abdominal subcutaneous and intrabdominal omental adipose tissue were obtained from men and women who underwent laparoscopic bariatric surgery.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- gender: Paired samples of abdominal subcutaneous and intrabdominal omental adipose tissue were obtained from men and women who underwent bariatric surgery.
  Interventions: Genetic: gender

INTERVENTIONS:
Genetic: gender — Paired samples of abdominal subcutaneous and intrabdominal omental adipose tissue were obtained from men and women who underwent bariatric surgery.
  Other Names: BMI were all over 40 kg/ m2

SUMMARY:
To investigate:

1. Associations between miRNA and insulin signaling-related gene expressions in abdominal adipose tissues in obese subjects.
2. Differences in miRNAs expressed by intrabdominal omental adipose tissues between genders.

DETAILED DESCRIPTION:
Compared the differences in microRNA expressions of abdominal adipose tissue in morbid obese male and female subjects to elucidate the possible regulatory role of microRNA in insulin signaling-related gene expression levels and its association with biochemical markers. We hope to find a miRNA that can be used to predict the syndrome associated with obesity.

ELIGIBILITY:
Inclusion Criteria:

* Morbid obesity,BMIs> 40 kg/m2
* Subjects who underwent bariatric surgery

Exclusion Criteria:

* Obese subjects with complicated metabolic disorders
* Thyroid disease

Ages: 19 Years to 63 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Paired samples of abdominal subcutaneous and intrabdominal omental adipose tissue were obtained from men (n = 9) and women (n =10) who underwent bariatric surgery. Their BMI were all over 40 kg/ m2, and ages between 19-63 years.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-06; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
MicroRNA expression in abdominal omental adipose tissues | up to 28 weeks
  MicroRNA-125a-3p expression in abdominal omental adipose tissues is associated with insulin signaling-related gene expression levels in morbid obesity

CONTACTS AND LOCATIONS:
Overall Officials: Wang Weu, Study Director — Comprehensive Weight Management Center Taipei Medical University Hospital
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan, Taiwan

REFERENCES:
- [Background] Brennecke J, Stark A, Russell RB, Cohen SM. Principles of microRNA-target recognition. PLoS Biol. 2005 Mar;3(3):e85. doi: 10.1371/journal.pbio.0030085. PMID 15723116
- [Background] Bartel DP. MicroRNAs: genomics, biogenesis, mechanism, and function. Cell. 2004 Jan 23;116(2):281-97. doi: 10.1016/s0092-8674(04)00045-5. PMID 14744438
- [Background] Hilton C, Neville MJ, Karpe F. MicroRNAs in adipose tissue: their role in adipogenesis and obesity. Int J Obes (Lond). 2013 Mar;37(3):325-32. doi: 10.1038/ijo.2012.59. Epub 2012 Apr 24. PMID 22531086
- [Background] Krotkiewski M, Bjorntorp P, Sjostrom L, Smith U. Impact of obesity on metabolism in men and women. Importance of regional adipose tissue distribution. J Clin Invest. 1983 Sep;72(3):1150-62. doi: 10.1172/JCI111040. PMID 6350364
- [Result] Jiang L, Huang Q, Zhang S, Zhang Q, Chang J, Qiu X, Wang E. Hsa-miR-125a-3p and hsa-miR-125a-5p are downregulated in non-small cell lung cancer and have inverse effects on invasion and migration of lung cancer cells. BMC Cancer. 2010 Jun 22;10:318. doi: 10.1186/1471-2407-10-318. PMID 20569443
- [Result] Herrera BM, Lockstone HE, Taylor JM, Wills QF, Kaisaki PJ, Barrett A, Camps C, Fernandez C, Ragoussis J, Gauguier D, McCarthy MI, Lindgren CM. MicroRNA-125a is over-expressed in insulin target tissues in a spontaneous rat model of Type 2 Diabetes. BMC Med Genomics. 2009 Aug 18;2:54. doi: 10.1186/1755-8794-2-54. PMID 19689793
- [Result] John B, Enright AJ, Aravin A, Tuschl T, Sander C, Marks DS. Human MicroRNA targets. PLoS Biol. 2004 Nov;2(11):e363. doi: 10.1371/journal.pbio.0020363. Epub 2004 Oct 5. PMID 15502875
- [Result] Kanehisa M, Goto S. KEGG: kyoto encyclopedia of genes and genomes. Nucleic Acids Res. 2000 Jan 1;28(1):27-30. doi: 10.1093/nar/28.1.27. PMID 10592173
- [Result] Gustafson B. Adipose tissue, inflammation and atherosclerosis. J Atheroscler Thromb. 2010 Apr 30;17(4):332-41. doi: 10.5551/jat.3939. Epub 2010 Feb 3. PMID 20124732
- [Result] O'Connell J, Lynch L, Cawood TJ, Kwasnik A, Nolan N, Geoghegan J, McCormick A, O'Farrelly C, O'Shea D. The relationship of omental and subcutaneous adipocyte size to metabolic disease in severe obesity. PLoS One. 2010 Apr 1;5(4):e9997. doi: 10.1371/journal.pone.0009997. PMID 20376319
- [Result] Wellen KE, Hotamisligil GS. Inflammation, stress, and diabetes. J Clin Invest. 2005 May;115(5):1111-9. doi: 10.1172/JCI25102. PMID 15864338
- [Result] Niswender KD, Morrison CD, Clegg DJ, Olson R, Baskin DG, Myers MG Jr, Seeley RJ, Schwartz MW. Insulin activation of phosphatidylinositol 3-kinase in the hypothalamic arcuate nucleus: a key mediator of insulin-induced anorexia. Diabetes. 2003 Feb;52(2):227-31. doi: 10.2337/diabetes.52.2.227. PMID 12540590